CLINICAL TRIAL: NCT04896229
Title: Talk STEM Familia: Dual-Language Academic Vocabulary-Building Technology to Improve Educational, Career, and Health Outcomes Among Latinx Students
Brief Title: Talk STEM Familia: Dual-Language (TSFII)
Acronym: TSFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD013619-02; 5R44MD013619-03 (NIH)
Record Dates: First submitted 2020-10-29; First posted 2021-05-21 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Vocabulary Acquisition
Keywords: Dual language technology; scientific academic vocabulary

STUDY DESIGN:
Intervention Model Description: One intervention and two arms: Intervention and treatment-as-usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): Parent/student/dyads in the treatment condition will be sent program materials via mail and text or email, including smart-speaker hardware, wireless network bridges for wireless network connectivity, and web links to Talk STEM Familia, including set-up video tutorials, and graphic instructions. Intervention activities will take place in participants' homes over the 24-week intervention period and will include using the dual-language Talk STEM Familia technology to receive instruction, practice, and feedback on academic vocabulary.
  Interventions: Other: Talk STEM Familia Treatment Condition
- Treatment as usual (No Intervention): Parent/student dyads in this arm will receive treatment-as-usual (the vocabulary instruction regularly provided in their schools). They will receive the TSF technology after post-test data has been collected.

INTERVENTIONS:
Other: Talk STEM Familia Treatment Condition — This study has one intervention and two arms: experimental and treatment as usual. Participants randomized to the treatment condition will receive the TSF technology in addition to the vocabulary instruction, monitoring, or resources delivered by English Language Development programs (ELD) and schools. TSF will deliver frequent, brief, dual-language exercises to help families learn, practice and apply SAV words in conversation. Audio-visual lessons will support learning at all literacy levels, regardless of prior familiarity with STEM subjects. The complete TSF tool will contain approximately 72 minutes of video modeling and 12 hours of interactive exercises delivered over 24-weeks in brief, interactive, easy to assimilate lessons.
  Arms: Experimental: Intervention

SUMMARY:
The study will evaluate Talk STEM Familia (TSF) effects on student and parent scientific academic vocabulary knowledge and usage, scientific academic vocabulary (SAV) learning behaviors, academic self efficacy, and satisfaction with the program, including acceptance of the technology and its usability.

DETAILED DESCRIPTION:
The Investigators will work with research practice partners Lane Educational Services District (ESD) to disseminate bilingual electronic and printed recruitment materials to Latinx families in the elementary and middle schools throughout the 16 school districts in Lane County, OR. Recruitment materials will direct families to contact the project's bilingual staff by phone to receive study details and, following a brief screen, to engage in an informed consent process. 300 eligible Latinx English-learner parent/student dyads will be recruited. Students will be in grade 4-8; families will speak primarily Spanish in the home; and families will have a smartphone, tablet, or computer and Internet access at home.

The Investigators will administer the pre-test to all 300 parent/student dyads via Qualtrics and randomize 150 parent/student dyads to the TSF treatment, 150 parent/student dyads to the treatment-as-usual control condition. Each family will be assigned a non-identifiable user name linked only to their non-identifiable participant ID. The Investigators will then send the TSF program materials and links to the treatment group. These materials will include graphic and video tutorials on TSF set-up and use, including set-up of a wireless bridge that allows researchers to monitor the non-identifiable program usage. Bilingual telephone support will be provided during the 1-month set-up period and throughout the 24-week TSF intervention period. During the intervention, families in the treatment group will be asked to use TSF for 24 weeks. During that time, they will receive 3 notifications/week that prompt them to engage in program games and activities targeting 72 scientific academic vocabulary (SAV) words.

Half way through the 24-week intervention period, the Investigators will administer the mid-test via Qualtrics to all 300 parent/student dyads and following the 24-week intervention, the Investigators will administer the post-test via Qualtrics to all 300 parent/student dyads. Pre-, mid-, and post-test surveys will measure gains in knowledge and usage of the 72 SAV words TSF targets, academic self-efficacy, and academic enabling behaviors. Treatment group dyads will also complete a usability, technology acceptance, and consumer satisfaction survey at post-test. All 300 parent/student dyads will receive a smart speaker at pretest, and $100 at mid-test and post-test.

Following post-test, parent/student dyads in the treatment-as-usual control condition will receive TSF program materials.

ELIGIBILITY:
Inclusion Criteria:

1. Latinx English learner parent with a student (grade 4-8)
2. Speaking primarily Spanish in the home
3. Having a smartphone, tablet, or computer
4. Having Internet in the home
5. Being the student (grade 4-8) of a participating parent

Exclusion Criteria:

1. N/A

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apthorp, H., Randel, B., Cherasaro, T., Clark, T., McKeown, M., & Beck, I. (2012). Effects of a supplemental vocabulary program on word knowledge and passage comprehension. Journal of Research on Educational Effectiveness, 5, 160-188.
- [Background] Bandura A, Barbaranelli C, Caprara GV, Pastorelli C. Self-efficacy beliefs as shapers of children's aspirations and career trajectories. Child Dev. 2001 Jan-Feb;72(1):187-206. doi: 10.1111/1467-8624.00273. PMID 11280478
- [Background] Betts, J. E., Appleton, J. J., Reschly, A. L., Christenson, S. L., & Huebner, E. S. (2010). A study of the factorial invariance of the Student Engagement Instrument (SEI): Results from middle and high school students. School Psychology Quarterly, 25(2), 84-93.
- [Background] Davis, F. D., Jr. (1986). A technology acceptance model for empirically testing new end-user information systems: Theory and results (Doctoral dissertation, Massachusetts Institute of Technology). http://hdl.handle.net/1721.1/15192
- [Background] McKeown, M., Beck, I., Omanson, R., & Perfetti, C. (1983). The effects of long-term vocabulary instruction on reading comprehension: A replication. Journal of Reading Behavior, 15, 3-18.
- [Background] Beck, I. L., Perfetti, C. A., & McKeown, M. G. (1982). Effects of long-term vocabulary instruction on lexical access and reading comprehension. Journal of Educational Psychology, 74, 506-521.
- See also: McKeown, M., Beck, I., Omanson, R., & Perfetti, C. (1983). The effects of long-term vocabulary instruction on reading comprehension: A replication. Journal of Reading Behavior, 15, 3-18. — https://scholar.google.com/citations?user=cz3hqv4AAAAJ&hl=en
- See also: Davis, F. D., Jr. (1986). A technology acceptance model for empirically testing new end-user information systems: Theory and results (Doctoral dissertation, Massachusetts Institute of Technology). http://hdl.handle.net/1721.1/15192 — https://dspace.mit.edu/handle/1721.1/15192
- See also: Bandura A, Barbaranelli C, Caprara GV, Pastorelli C. Self-efficacy beliefs as shapers of children's aspirations and career trajectories. Child Dev. 2001 Jan-Feb;72(1):187-206. — https://www.uky.edu/~eushe2/Bandura/Bandura2001CD.pdf
- See also: Apthorp, H., Randel, B., Cherasaro, T., Clark, T., McKeown, M., & Beck, I. (2012). Effects of a supplemental vocabulary program on word knowledge and passage comprehension. Journal of Research on Educational Effectiveness, 5, 160-188. — https://eric.ed.gov/?id=EJ961442
- See also: Beck I, Perfetti C, Mckeown M, (1982). Effects of long-term vocabulary instruction on lexical access and reading comprehension. Journal of Education Psychology, 74(4): 506-521. doi:10.1037/0022-0663.74.4.506 — https://www.researchgate.net/publication/232540440_Effects_of_long-term_vocabulary_instruction_on_lexical_access_and_reading_comprehension

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 400 participants, however, only 168 parents and student dyads (N = 336) were randomized to the study. The remaining 64 participants were part of the formative research and were never meant to be part of the randomized study. In the Protocol Enrollment, the Number Started and Number Completed reflect dyads. See the Milestones for specificity at the parent and youth levels.
Period: Overall Study
Arm/Group | Experimental: Intervention | Treatment as Usual
Started | 164 | 172
Time 1: Parents | 82 | 86
Time1: Youth | 79 | 75
Time 2: Parents | 50 | 62
Time2: Youth | 46 | 56
Time3: Parent | 27 | 28
Time 3: Youth | 24 | 31
Completed | 51 | 59
Not Completed | 113 | 113
Not completed — Lost to Follow-up | 113 | 113

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 164 | 172 | 336
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 82 | 86 | 168
  Between 18 and 65 years | 81 | 86 | 167
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 131 | 246
  Male | 49 | 41 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 1 | 1 | 2
  White | 21 | 42 | 63
  More than one race | 114 | 111 | 225
  Unknown or Not Reported | 25 | 13 | 38
Relationship to Child [Count of Participants; unit: Participants] — The parents relationsihp to the child participating in the study.
  Participants
    Parent report - Daughter | 45 | 45 | 90
    Parent report - Son | 38 | 35 | 73
    Parent report - Other | 1 | 0 | 1
    NA for child or missing parent report | 80 | 92 | 172

OUTCOME MEASURES:

1. Primary Outcome: Student Scientific Academic Vocabulary (SAV) Word Meaning (AVM)
Description: AVM (Academic Vocabulary Meaning) will measure change in student vocabulary knowledge (multiple choice test of meaning). The multiple choice test is based on the assessment used in Beck et al. (1982) and McKeown et al. (1983) with middle school students. Scores were computed as the total percentage of vocabulary words correctly identified out of 72. Score could range from 0 to 100 and higher scores indicate greater levels of vocabulary knowledge.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: percentage of vocabulary words correct
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
percentage of vocabulary words correct
  T1 | 60.63 (17.42) | 62.43 (18.27)
  T2 | 65.82 (19.34) | 67.35 (15.97)
  T3 | 69.79 (17.21) | 61.80 (23.37)
Statistical Analysis 1: Comparison: Experimental: Intervention; The results show the condition x time interaction from the growth model, and the parameter estimate describes the relative change of the intervention condition to the treatment-as-usual condition, for a unit change in time; Test type: Superiority; p = .022, t-test, 2 sided; Slope = 1.20, Standard Error of Mean 0.52

2. Primary Outcome: Parent SAV Word Meaning (AVM)
Description: AVM (Academic Vocabulary Meaning) will measure change in parent vocabulary knowledge (multiple choice test of meaning). The multiple choice test is based on the assessment used in Beck et al. (1982) and McKeown et al. (1983) with middle school students. Scores were computed as the total percentage of vocabulary words correctly identified out of 72. Score could range from 0 to 100 and higher scores indicate greater levels of vocabulary knowledge.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: percentage of vocabulary words correct
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 82 | 86
percentage of vocabulary words correct
  T1 | 72.27 (13.20) | 72.53 (11.78)
  T2 | 75.49 (14.90) | 73.20 (14.93)
  T3 | 76.90 (15.20) | 76.30 (11.46)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .800, t-test, 2 sided; Slope = 0.09, Standard Error of Mean 0.35

3. Primary Outcome: Student SAV Word Usage (AVWU)
Description: AVMU (Academic Vocabulary Meaning Usage) will measure change in student ability to correctly use vocabulary words in sentence contexts. The sentence verification test is similar to the Test of Instructed Word Knowledge in Vocabulary used in the Apthorp et al. (2012) study of vocabulary learning in middle school. Scores were computed as the total percentage of vocabulary words correctly used in sentence context out of 72 items. Score could range from 0 to 100 and higher scores indicate greater levels of vocabulary words used correctly in a sentence.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: percentage of words used correctly
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
percentage of words used correctly
  T1 | 71.04 (14.31) | 72.05 (12.44)
  T2 | 74.27 (15.94) | 72.94 (13.90)
  T3 | 76.50 (12.11) | 70.93 (17.76)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .235, t-test, 2 sided; Slope = 0.58, Standard Error of Mean 0.49

4. Primary Outcome: Parent SAV Word Usage (AVWU)
Description: AVMU (Academic Vocabulary Meaning Usage) will measure change in parent ability to correctly use vocabulary words in sentence contexts. The sentence verification test is similar to the Test of Instructed Word Knowledge in Vocabulary used in the Apthorp et al. (2012) study of vocabulary learning in middle school. Scores were computed as the total percentage of vocabulary words correctly used in sentence context out of 72 items. Score could range from 0 to 100 and higher scores indicate greater levels of vocabulary words used correctly in a sentence.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: percentage of words used correctly
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 82 | 86
percentage of words used correctly
  T1 | 80.84 (11.19) | 80.59 (10.34)
  T2 | 82.38 (8.59) | 79.98 (12.33)
  T3 | 82.41 (10.43) | 79.90 (9.42)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .325, t-test, 2 sided; Slope = 0.29, Standard Error of Mean 0.30

5. Secondary Outcome: Student Use of SAV: AVUB
Description: AVUB (Academic Vocabulary Usage Behaviors) will measure change in student use of SAV words (10 items). Items were adapted from: the Student Engagement Instrument (SEI; Betts, Appleton, Reschly, et al., 2010). Items used a 4-point response option (1 = not at all, 4 = 3-4 times per week) and a mean score was computed (alpha = .89) and could range from 1 to 4. Higher scores indicated greater use of SAV words.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
score on a scale
  T1 | 2.27 (0.67) | 2.26 (0.73)
  T2 | 2.43 (0.72) | 2.40 (0.69)
  T3 | 2.28 (0.64) | 2.42 (0.80)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .502, t-test, 2 sided; Slope = -0.02, Standard Error of Mean 0.03

6. Secondary Outcome: Parent Use of SAV: AVUB
Description: AVUB (Academic Vocabulary Usage Behaviors) will measure change in parent use of SAV words (10 items). Items were adapted from: the Student Engagement Instrument (SEI; Betts, Appleton, Reschly, et al., 2010). Items used a 4-point response option (1 = not at all, 4 = 3-4 times per week) and a mean score was computed (alpha = .91) and could range from 1 to 4. Higher scores indicated greater use of SAV words.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 82 | 86
score on a scale
  T1 | 1.78 (0.63) | 1.84 (0.75)
  T2 | 2.38 (0.62) | 2.02 (0.74)
  T3 | 2.46 (0.67) | 2.14 (0.72)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .005, t-test, 2 sided; Slope = 0.06, Standard Error of Mean 0.02

7. Secondary Outcome: Student Confidence in Using SAV Words (AVC)
Description: AVC will measure student confidence in using SAV words (10 items). Items were adapted from the Efficacy to Influence School-related Performance subscale of the Parental Self-Efficacy Scale (PSES; Bandura, et al., 2001). Items were developed using procedures for developing self-efficacy scales (Bandura et al., 2001). Items used a 5-point response option (1 = not at all confident, 5 = extremely confident) and a mean score was computed (alpha = .89) and could range from 1 to 5. Higher scores indicated greater confidence using SAV words.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
score on a scale
  T1 | 2.82 (0.84) | 2.77 (0.83)
  T2 | 2.99 (1.00) | 2.76 (1.04)
  T3 | 3.04 (0.73) | 3.05 (1.15)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .712, t-test, 2 sided; Slope = -0.10, Standard Error of Mean 0.03

8. Secondary Outcome: Parent Confidence in Using SAV Words (AVC)
Description: AVC will measure parent confidence in using SAV words (10 items). Items were adapted from the Efficacy to Influence School-related Performance subscale of the Parental Self-Efficacy Scale (PSES; Bandura, et al., 2001). Items were developed using procedures for developing self-efficacy scales (Bandura et al., 2001). Items used a 5-point response option (1 = not at all confident, 5 = extremely confident) and a mean score was computed (alpha = .95) and could range from 1 to 5. Higher scores indicated greater confidence using SAV words.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 82 | 86
score on a scale
  T1 | 2.72 (0.94) | 2.69 (0.97)
  T2 | 2.73 (0.85) | 2.60 (0.89)
  T3 | 2.78 (1.07) | 2.78 (1.07)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .245, t-test, 2 sided; Slope = 0.03, Standard Error of Mean 0.03

9. Secondary Outcome: Student Interest in Choosing STEM Careers (STEM)
Description: STEM will measure student interest in choosing STEM careers (4 items). Items were adapted from: the Student Engagement Instrument (SEI; Betts, Appleton, Reschly, et al., 2010) and the Efficacy to Influence School-related Performance subscale of the Parental Self-Efficacy Scale (PSES; Bandura, et al., 2001). Items used a 5-point response option (1 = not at all interested, 5 = extremely interested) and a mean score was computed (alpha = .69) and could range from 1 to 5. Higher scores indicated greater interest using SAV words.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
score on a scale
  T1 | 3.13 (0.74) | 3.08 (0.83)
  T2 | 3.04 (0.90) | 2.98 (1.00)
  T3 | 2.94 (0.83) | 3.12 (0.98)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .282, t-test, 2 sided; Slope = -0.03, Standard Error of Mean 0.03

10. Secondary Outcome: Parent Academic Support (AEB)
Description: AEB will measure parent academic support behaviors (20 items). Efficacy to Influence School-related Performance subscale of the Parental Self-Efficacy Scale (PSES; Bandura, et al., 2001). Items used a 9-point response option (1 = nothing, 9 = a great deal) and a mean score was computed (alpha = .94) and could range from 1 to 9. Higher scores indicated greater efficacy to influence school performance.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 82 | 86
score on a scale
  T1 | 7.15 (1.50) | 7.37 (1.39)
  T2 | 7.34 (1.37) | 7.49 (1.33)
  T3 | 7.27 (1.27) | 7.20 (1.37)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .289, t-test, 2 sided; Slope = 0.04, Standard Error of Mean 0.03

11. Secondary Outcome: Student Academic Learning (ALB)
Description: ALB will measure student academic learning behaviors (20 items). Items used a 5-point response option (1 = strongly disagree, 5 = strongly agree) and a mean score was computed (alpha = .90) and could range from 1 to 5. Higher scores indicated greater levels of perceived academic learning behaviors.
Time Frame: Baseline, 12 weeks (mid-treatment), and 24 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Intervention | Treatment as Usual
Number analyzed (Participants) | 79 | 75
score on a scale
  T1 | 4.16 (0.48) | 4.13 (0.54)
  T2 | 4.00 (0.67) | 4.15 (0.57)
  T3 | 3.93 (0.56) | 4.04 (0.87)
Statistical Analysis 1: Comparison: Experimental: Intervention vs Treatment as Usual; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .296, t-test, 2 sided; Slope = -0.02, Standard Error of Mean 0.02

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from after receipt of the consent form through study completion, an average of 6-months
Arm/Group | Experimental: Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/172
Other Adverse Events (participants affected / at risk) | 0/164 | 0/172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04896229/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04896229/ICF_001.pdf